CLINICAL TRIAL: NCT00414180
Title: Bupropion SR for Treating Smokeless Tobacco Use
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: West Virginia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-007293; R01 9088
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Smokeless Tobacco
MeSH Terms: conditions — Tobacco Use

INTERVENTIONS:
Drug: Bupropion SR

SUMMARY:
To determine the efficacy and safety of bupropion SR for quitting tobacco in smokeless tobacco users.

DETAILED DESCRIPTION:
CONTEXT: No pharmacotherapies have been shown to increase long-term (≥ 6 month) tobacco abstinence rates among smokeless tobacco (ST) users, although bupropion SR has demonstrated potential efficacy in pilot studies.

OBJECTIVE: To determine the efficacy and safety of bupropion SR for tobacco abstinence among ST users compared with placebo.

DESIGN, SETTING, AND PARTICIPANTS: A randomized, double-blind, placebo-controlled trial conducted between August 2003 to May 2005 at two research centers with a 12-week treatment period and follow-up of smoking status to week 52.

INTERVENTION: Bupropion SR titrated to 150 mg twice daily or placebo for 12 weeks plus weekly behavioral interventions.

Main Outcome Measures: The primary endpoint was 7-day point-prevalence tobacco abstinence rate at week 12. Secondary outcomes included the prolonged and continuous tobacco abstinence rates at weeks 12, 24, and 52.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* used ST daily for at least one year
* in good general health
* willing to complete all study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225
Dates: Start 2003-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
7-day point-prevalence tobacco abstinence rate at week 12

SECONDARY OUTCOMES:
prolonged and continuous tobacco abstinence rates at weeks 12, 24, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Lowell C. Dale, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States